CLINICAL TRIAL: NCT03066011
Title: Observational Disease Registry of Patients Treated With Systemic Mold-Active Triazoles
Brief Title: Registry of Patients Treated With Systemic Mold-Active Triazoles
Status: Completed | Type: Observational
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Other Study IDs: 9766-MA-3034
Record Dates: First submitted 2017-02-23; First posted 2017-02-28 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2020-08

CONDITIONS: Invasive Fungal Infection
Keywords: mold-active triazoles
MeSH Terms: conditions — Invasive Fungal Infections | interventions — isavuconazole; Voriconazole; posaconazole

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Isavuconazonium sulfate Group: Oral and Intravenous
  Interventions: Drug: Isavuconazonium sulfate
- Voriconazole Group: Oral and Intravenous
  Interventions: Drug: Voriconazole
- Posaconazole Group: Oral and Intravenous
  Interventions: Drug: Posaconazole

INTERVENTIONS:
Drug: Isavuconazonium sulfate — Oral and Intravenous
  Other Names: Cresemba
  Groups: Isavuconazonium sulfate Group
Drug: Voriconazole — Oral and Intravenous
  Other Names: Vfend
  Groups: Voriconazole Group
Drug: Posaconazole — Oral and intravenous
  Other Names: Noxafil
  Groups: Posaconazole Group

SUMMARY:
The purpose of this study is to describe representative real-world patterns of care for the management of invasive fungal infections (IFIs), including invasive mold infection (IMI). Specifically, the study goals are to examine real world patient characteristics and treatment patterns, associated healthcare resource utilization, and outcomes associated with use of mold-active triazoles (MATs) to treat invasive fungal infections (IFIs).

ELIGIBILITY:
Inclusion Criteria:

* Patients taking one of the following target drugs at the time of enrollment: isavuconazonium sulfate (ISAV), voriconazole (VORI), posaconazole (POSA).

Exclusion Criteria:

* Currently enrolled in any clinical trial with an investigational antifungal agent. Individuals who subsequently enroll in an investigational antifungal study will be discontinued and data collected up to the time of investigational product will be evaluable.
* Patients who died before entering the study.
* Patients who previously participated in this registry.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients on a mold-active triazole
Sampling Method: Probability Sample
Enrollment: 2015 (Actual)
Dates: Start 2017-03-16 (Actual); Primary Completion 2020-04-24 (Actual); Study Completion 2020-04-24 (Actual)

PRIMARY OUTCOMES:
Treatment patterns of care assessed by reason for therapy | 5 years
  Assessments of patient patterns of care will be summarized by MAT treatment at baseline and overall.
Treatment patterns of care assessed by category of diagnosis at time of therapy initiation | 5 years
  Assessments of patient patterns of care will be summarized by MAT treatment at baseline and overall.
Treatment patterns of care assessed by onset of treatment/prophylaxis | 5 years
  Assessments of patient patterns of care will be summarized by MAT treatment at baseline and overall.
Treatment patterns of care assessed by length of treatment/prophylaxis | 5 years
  Assessments of patient patterns of care will be summarized by MAT treatment at baseline and overall.
Treatment patterns of care assessed by use of diagnostic method(s) | 5 years
  Assessments of patient patterns of care will be summarized by MAT treatment at baseline and overall.
Treatment patterns of care assessed by type of diagnostic method(s) used | 5 years
  Assessments of patient patterns of care will be summarized by MAT treatment at baseline and overall.
Treatment patterns of care assessed by use of therapeutic drug monitoring (TDM) | 5 years
  Assessments of patient patterns of care will be summarized by MAT treatment at baseline and overall.
Treatment patterns of care assessed by occurrence of drug-drug interactions (DDI) | 5 years
  Assessments of patient patterns of care will be summarized by MAT treatment at baseline and overall.
Treatment patterns of care assessed by the sequence of invasive fungal infection treatment (IFI) | 5 years
  Assessments of patient patterns of care will be summarized by MAT treatment at baseline and overall.
Treatment patterns of care assessed by discontinuation due to adverse events (AEs) or other reasons | 5 years
  Assessments of patient patterns of care will be summarized by MAT treatment at baseline and overall.
Patient characteristics assessed by underlying host/risk factors | 5 years
  The summaries of patient characteristics will be by MAT treatment at baseline and overall.
Patient characteristics assessed by patient baseline characteristics | 5 years
  The summaries of patient characteristics will be by MAT treatment at baseline and overall.
Patient characteristics assessed by fungal disease diagnosis | 5 years
  The summaries of patient characteristics will be by MAT treatment at baseline and overall.
Patient characteristics assessed by pathogen treated | 5 years
  The summaries of patient characteristics will be by MAT treatment at baseline and overall.
Patient characteristics assessed by pathogen susceptibility | 5 years
  The summaries of patient characteristics will be by MAT treatment at baseline and overall.
Patient characteristics assessed by site of fungal infection | 5 years
  The summaries of patient characteristics will be by MAT treatment at baseline and overall.

SECONDARY OUTCOMES:
Overall healthcare resource utilization assessed by hospitalization length of stay (LOS) | 5 years
  Assessments of overall healthcare resource inpatient utilization will be summarized
Overall healthcare resource utilization assessed by time spent in Intensive Care Unit (ICU) | 5 years
  Assessments of overall healthcare resource inpatient utilization will be summarized
Overall healthcare resource utilization assessed by time spent on ventilator in ICU | 5 years
  Assessments of overall healthcare resource inpatient utilization will be summarized
Overall healthcare resource utilization assessed by number of additional fungal specific diagnostics and interventions after MAT initiation | 5 years
  Assessments of overall healthcare resource inpatient utilization will be summarized
Overall healthcare resource utilization assessed by frequency of therapeutic drug monitoring (TDM) | 5 years
  Assessments of overall healthcare resource inpatient utilization will be summarized
Overall healthcare resource utilization assessed by incidence of discharge to a skilled nursing facility (SNF) or long term care (LTC) facility | 5 years
  Assessments of overall healthcare resource inpatient utilization will be summarized
Overall healthcare resource utilization assessed by length of stay at SNF or LTC facility | 5 years
  Assessments of overall healthcare resource inpatient utilization will be summarized
Overall healthcare resource utilization assessed by reason for admission to SNF or LTC facility | 5 years
  Assessments of overall healthcare resource inpatient utilization will be summarized
Overall healthcare resource utilization assessed by incidence of hospital readmissions at 30 and 90 days within a 5-year period | 5 years
  Assessments of overall healthcare resource inpatient utilization will be summarized
Overall healthcare resource utilization assessed by duration of hospital readmissions at 30 and 90 days within a 5-year period | 5 years
  Assessments of overall healthcare resource inpatient utilization will be summarized
Overall healthcare resource utilization assessed by outpatient utilization | 5 years
  Number of ED visits during the follow-up period
Overall healthcare resource utilization assessed by frequency of outpatient visits within 30 and 90 days within a 5-year period | 5 years
  Assessments of overall healthcare resource outpatient utilization will be summarized
Overall healthcare resource utilization assessed by primary reason for outpatient office visits within 30 and 90 days within a 5-year period | 5 years
  Assessments of overall healthcare resource outpatient utilization will be summarized

CONTACTS AND LOCATIONS:
Overall Officials: Senior Medical Director, Study Director — Astellas Pharma Global Development, Inc.
Locations (56):
- United States (56):
  - University of Alabama - Birmingham, Birmingham, Alabama
  - St. Joseph's Hospital, Phoenix, Arizona
  - Mayo Clinic, Phoenix, Arizona
  - University of Arizona, Tucson, Arizona
  - University of California, Davis, California
  - David Geffen School of Medicine, Los Angeles, California
  - Stanford Health Care, Palo Alto, California
  - Olive View UCLA Medical Center, Sylmar, California
  - LA BioMed, Torrance, California
  - University of Colorado, Aurora, Colorado
  - Yale School of Medicine, New Haven, Connecticut
  - Emory University, Atlanta, Georgia
  - Augusta University, Augusta, Georgia
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Northwestern University, Chicago, Illinois
  - University of Illinois at Chicago, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Loyola University, Chicago, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Indiana University Health, Indianapolis, Indiana
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Kentucky, Lexington, Kentucky
  - Norton Cancer Institute, Louisville, Kentucky
  - Tulane Medical Center, New Orleans, Louisiana
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Michigan Cancer Center, Ann Arbor, Michigan
  - Wayne State University, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Children's Mercy Hospital, Kansas City, Missouri
  - Washington University St. Louis, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Cooper University Hospital, Camden, New Jersey
  - Robert Wood Johnson University Hospital Somerset, Somerville, New Jersey
  - Roswell Park Cancer Center, Buffalo, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Weill Cornell Medicine of Cornell University and New York Presbyterian Hospital, New York, New York
  - Duke University, Durham, North Carolina
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
  - Case Western Reserve University, Cleveland, Ohio
  - Regional Infectious Disease and Infusion Center, Inc., Lima, Ohio
  - Good Samaritan Hospital, Corvallis, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Drexel University College of Medicine, Philadelphia, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - St. Jude Childrens Research Hospital, Memphis, Tennessee
  - University of Texas Health Science Center, Houston, Texas
  - Virginia Commonwealth University, Richmond, Virginia
  - Swedish Health System, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington
  - WVU Medicine, Morgantown, West Virginia

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.